CLINICAL TRIAL: NCT03034031
Title: Classifying Neuro-imaging Measures Predicting Rehabilitation Outcome Following Pediatric Closed Head Injuries.
Brief Title: MR Imaging Study of TBI in Children
Acronym: MISTIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Abigail livny-ezer, Head of functional neuromaging lab, Department of Diagnostic Imaging, Sheba Medical Center
Other Study IDs: 3211-16-SMC
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: Traumatic Brain Injury; Children; Pediatric; MRI; fMRI; Cognition; DTI; Longitudinal; Connectivity; DAI; Neuropsychology; Rehabilitation
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project will combine the data collected from structural and functional MRI scans and neuropsychology performance post-TBI in children. Patients will be followed for a year, in order to examine the brain and cognitive recovery post head injury.

DETAILED DESCRIPTION:
Traumatic brain injury in childhood has an cumulative effect that leads to impairments in cognitive functions such as deficits in memory, executive functions and attention. The cognitive impairment is the main cause of disabilities in the injured population, and has a different effect depending on the type and severity of the injury.

Imaging after brain trauma serves as a useful diagnostic tool in identifying the head trauma's results. Therefore, in recent years, using imaging methods, studies have tried to find measures which will be able to predict the functional outcome after brain injury in children, and assist in developing a personalized rehabilitation program. The combination of advanced imaging techniques with neuropsychological assessment within the early stage of the injury and during a year of followup, will allow us to establish the relationship between those measures and the functional recovery result of the children. This multi-analysis will enable us to have a deeper understanding of the neuroplasticity process and the functional recovery after brain injury in the developing young brain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 9-18 years old, which are/were hospitalized in the Pediatric Rehabilitation Department, Sheba Medical Center
2. Glasgow coma scale score of 3-15.
3. Hebrew as mother-tongue

Exclusion Criteria:

1. History of neurological disorders, mental retardation or a previous head injury.
2. Current diagnosis or history of psychiatric disorders.
3. Cardiovascular instability.
4. Metabolic instability (water, electrolytes, sugar).
5. Fever or evidence of microbiological pollutant.
6. Uncontrolled seizures. 7 . Hydrocephalus.

8. Deafness or blindness. 9. Renal failure.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: study population will include 1 group of subjects: group 1: young subjects, age 9-18, after traumatic brain injury
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-06-24 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Functional MRI | 12 months
  fMRI brain activation to a cognitive tasks
Structural MRI | 12 months
  MRI Structural changes using different methods
neuropsychological tests | 12 months
  Cognitive scores on neuropsychological testing

SECONDARY OUTCOMES:
Associations between the cognitive performance and the imaging methods | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Livny-Ezer, PhD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center Tel Hashomer, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Livny A, Biegon A, Kushnir T, Harnof S, Hoffmann C, Fruchter E, Weiser M. Cognitive Deficits Post-Traumatic Brain Injury and Their Association with Injury Severity and Gray Matter Volumes. J Neurotrauma. 2017 Apr 1;34(7):1466-1472. doi: 10.1089/neu.2016.4598. Epub 2016 Dec 2. PMID 27750571
- [Background] Anderson VA, Anderson P, Northam E, Jacobs R, Mikiewicz O. Relationships between cognitive and behavioral measures of executive function in children with brain disease. Child Neuropsychol. 2002 Dec;8(4):231-40. doi: 10.1076/chin.8.4.231.13509. PMID 12759820
- [Background] Anderson V, Catroppa C. Recovery of executive skills following paediatric traumatic brain injury (TBI): a 2 year follow-up. Brain Inj. 2005 Jun;19(6):459-70. doi: 10.1080/02699050400004823. PMID 16101268
- [Background] Anderson V, Catroppa C, Morse S, Haritou F, Rosenfeld J. Recovery of intellectual ability following traumatic brain injury in childhood: impact of injury severity and age at injury. Pediatr Neurosurg. 2000 Jun;32(6):282-90. doi: 10.1159/000028956. PMID 10971189
- [Background] Keightley ML, Sinopoli KJ, Davis KD, Mikulis DJ, Wennberg R, Tartaglia MC, Chen JK, Tator CH. Is there evidence for neurodegenerative change following traumatic brain injury in children and youth? A scoping review. Front Hum Neurosci. 2014 Mar 19;8:139. doi: 10.3389/fnhum.2014.00139. eCollection 2014. PMID 24678292